CLINICAL TRIAL: NCT07200960
Title: Analgesic Efficacy of Erector Spinae Plane Block Versus Retrolaminar Block in Patients Undergoing Major Oncological Breast Surgery: a Randomized Controllled Trial
Brief Title: ESP vs Retrolaminar Block: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-23-02
Record Dates: First submitted 2025-09-29; First posted 2025-10-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Pain Management; Opoid Managment
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: will be asked regarding the group of blocks being employed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient receiving ESPB for major oncological breast surgery (Experimental): Patient receiving ESPB for major oncological breast surgery
  Interventions: Procedure: ESPB
- Patient receiving Retrolaminar block for major oncological breast surgery (Experimental): Patient receiving ESPB for major oncological breast surgery
  Interventions: Procedure: ESPB

INTERVENTIONS:
Procedure: ESPB — Patient receiving ESPB for major oncological breast surgery Patient receiving Retrolaminar Block for major oncological breast surgery
  Other Names: Retrolaminar Block

SUMMARY:
The study aims to compare the efficacy in pain control and total opioid consumption after the use of ESPB and retrolaminar block in patients undergoing major oncological breast surgery..

DETAILED DESCRIPTION:
The study aims to compare the efficacy in pain control and total opioid consumption after the use of ESPB and retrolaminar block in patients undergoing major oncological breast surgery..

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 18- 60 years ASA 1 and 2

Exclusion Criteria:

* Patient refusal Allergic reaction infection emergency case BMI >35

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female population has a bigger incision as compared to male population.
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pain score of patients receiving ESPB and retrolaminar block | 2hours post surgery
  Numeric rating scale score

SECONDARY OUTCOMES:
Comparison of total opioid consumption in 24 hours of patients receiving ESPB and retrolaminar block | 24 hours post surgery
  total consumption of opioids in MG

CONTACTS AND LOCATIONS:
Locations (1):
- Shaukat Khanum Memorial Cancer Hospital & Research Centre., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No